CLINICAL TRIAL: NCT06191354
Title: A Multicenter, Open, Dose-escalation Clinical Study Evaluating the Safety, Initial Efficacy, and Immunogenicity of SKG0201 Injection in Patients With Spinal Muscular Atrophy Type 1
Brief Title: A Clinical Study Evaluating the Safety and Efficacy of SKG0201 Injection in Patients With Spinal Muscular Atrophy Type 1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kun Sun (Other)
Responsible Party: Sponsor-Investigator, Kun Sun, Professor of Department of Pediatric Cardiology, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKG0201-001
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Spinal Muscular Atrophy 1
Keywords: SMA 1
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-escalation (Experimental): SKG0201 one-time deliver
  Interventions: Genetic: SKG0201 Injection

INTERVENTIONS:
Genetic: SKG0201 Injection — SKG0201 is a recombinant adeno-associated virus (rAAV) vector-based in vivo gene therapeutic product.
  Other Names: SKG0201

SUMMARY:
This is a clinical study to evaluate the safety and efficacy of gene therapy drug SKG0201 Injection in patients with spinal muscular atrophy Type 1 (SMA 1).

DETAILED DESCRIPTION:
This is a multicenter, open, dose-escalation clinical study to evaluate the safety, initial efficacy, and immunogenicity of SKG0201 injection in patients with spinal muscular atrophy type 1 (SMA 1).

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 SMA, defined by bi-allelic mutations in the SMN1 gene.
2. Age 180 days or younger at day of infusion.
3. Clinical history and signs are consistent with type I SMA, that is hypotonia on clinical examination, with delay in motor skills, poor head control, rounded shoulder posture, and joint hypermobility.
4. The legal guardian of the subject understands the purpose of the study, the possible risks and rights of the study, agrees that the subject can participate in the study, complete all research steps, tests and visits, and sign the ICF voluntarily.
5. During the study period, according to the change of the subject's condition, the subject's legal guardian is willing to perform standard treatment requirements as suggested by the researcher.

Exclusion Criteria:

1. Pulse oximetry < 96% saturation at screening while the patient is awake or asleep without any supplemental oxygen or respiratory support.
2. Weight-for-age below the 3rd percentile for the same sex and age based on WHO Child Growth Standards (WHO 2006).
3. Active viral infection with significant signs or symptoms and require systematic hospitalization.
4. In the presence of other severe infections or diseases.
5. Known allergy to prednisolone, other glucocorticoids, or their excipients.
6. Clinically significant abnormal laboratory values prior to administration.
7. Previously used other SMA drugs (such as Spinraza, Evrysdi, Zolgensma, etc.) or participated in clinical studies of other SMA drugs.
8. Had received previous or anticipated major surgical procedures during the study assessment period.

Max Age: 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2023-06-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs and SAEs | 18 months of age
  AEs: adverse events; SAEs: serious Adverse events
Incidence and characteristics of DLT | 4 weeks
  DLT: dose-limiting toxicity

SECONDARY OUTCOMES:
Survival rate | 14 months of age
  Survival is defined as avoidance of either death or permanent ventilation.
CHOP-INTEND score changes from baseline | 24 weeks
  CHOP-INTEND (Children's hospital of Philadelphia Infant Test of Neuromuscular Disorders) score ranges from 0 to 64 with higher scores indicating higher motor function.
Proportion of subjects who achieve developmental milestones with improvement in exercise intensity and function assessed according to BSID-III | 24 weeks
  Developmental milestones are defined according to BSID-III (Bayley Scales of Infant and Toddler Development Third Edition) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Sun, Doctor, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine; Yongguo Yu, Doctor, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (3):
- China (3):
  - West China Sencond Hospital, Sichuan University / West China women's and children's Hospital, Chengdu, Sichuan
  - Xinhua Hospital Affiliated To Shanghai Jiao Tong University School Of Medicine, Shanghai
  - National Children's Medical Center, Children's Hospital of Fudan University, Shanghai